CLINICAL TRIAL: NCT05608421
Title: 1MoreStep: Pilot Trial of an Intervention to Increase HIV Care Engagement and Reduce Intimate Partner Violence Among Black Women Living With HIV
Brief Title: 1MoreStep: An Intervention to Increase HIV Care Engagement and Reduce Intimate Partner Violence Among Black Women Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00350026; R34MH124586-01A1 (NIH)
Record Dates: First submitted 2022-10-31; First posted 2022-11-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Violence, Domestic; HIV; Stigma, Social; Engagement, Patient; Medication Adherence
Keywords: HIV; Intimate Partner Violence (IPV); Black women; Cognitive behavioral approach; Randomized Control Trial (RCT)
MeSH Terms: conditions — Social Stigma; Patient Participation; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of the two groups for the duration of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1MoreStep Intervention (Experimental): The intervention arm is 8 sessions (7 group and one individual) that meet weekly with a community health educator who is a Black woman and has experience implementing prior behavioral interventions with people who have experienced trauma and/or are LWH.
  Interventions: Behavioral: 1MoreStep
- Equal Attention Control (Active Comparator): The Equal Attention Control consists of 8 sessions (7 group and one individual) that meet weekly for 60-90 minutes. The control sessions provide equal attention and psychotherapeutic experience of a support group where participants can address issues important in their lives.
  Interventions: Behavioral: 1MoreStepControl

INTERVENTIONS:
Behavioral: 1MoreStep — Cognitive behavioral intervention to reduce HIV and IPV stigma.
  Arms: 1MoreStep Intervention
Behavioral: 1MoreStepControl — This is an equal attention control group.
  Arms: Equal Attention Control

SUMMARY:
This study tests a 5-session cognitive behavioral approach program (herein referred to as the 1MoreStep intervention) to train Black women living with HIV (BWLWHI) and exposed to intimate partner violence (IPV) in the past 2 years (hereafter, BWLWHI) in: 1) cognitive and behavioral skills to access internal and external sources of strength (e.g. self-reliance, safety net); safety strategies, knowledge about Undetectable = Untransmissible (U=U) and HIV care; and reduce internalized and anticipated stigma; 2) communication skills to respond to enacted HIV and IPV stigma and enlist social support; and 3) addressing structural barriers to HIV care engagement with an HIV navigator component. The intervention is informed by the HIV-Stigma Framework and a resilient-reintegration model which views women as active participants in responding to IPV and managing life with HIV.

Aim 1: Examine preliminary efficacy of the 1MoreStep intervention on: (a) IPV safety strategies (informal and formal resources, safety planning, and placating strategies at baseline, 3-month and 6-month follow-up visits); and (b) HIV care engagement (medical record confirmed visit with an HIV care provider, antiretroviral therapy (ART) prescription, medication adherence, and viral load status during 3-month and 6-month follow-up visits).

Aim 2: Examine the acceptability and feasibility of the 1MoreStep intervention operationalized by (a) quantitative measures: session attendance and fidelity to key intervention components and (b) qualitative interviews to assess: program fit, facilitators and barriers to participation, and using 1MoreStep intervention skills.

DETAILED DESCRIPTION:
HIV care engagement is essential to optimize the health of Black women LWH. Black women LWH have poorer health outcomes due to exposures to poverty, substance use, and violence as well as constrained support resources derived from historically unjust social policies. Baltimore City has the highest prevalence rates of HIV in Maryland. In 2018, nearly 1 in 5 (18.7%) people living with HIV, the majority of whom are Black, were not engaged in HIV care and only two-thirds had achieved viral suppression. Two critical aspects of HIV care engagement include at least two HIV care visits in a 12-month period 90 days apart and a prescription for ART as early as possible after HIV diagnosis. HIV care engagement among Black women LWH can be challenging; and exposure to IPV is a well-established barrier.

Black women LWH experience high rates of IPV victimization. Approximately 1 in 2 Black women report lifetime experiences of IPV compared to 1 in 3 White women. Women LWH and experiencing IPV are more likely to have a lower Clusters of differentiation 4(CD4) count and higher viral load; and delayed care poses heightened risks for ongoing HIV transmission in communities. Black women LWH also report higher rates of severe IPV, greater IPV frequency, and are more likely to be murdered by an abusive partner in the United States. Despite these stressors, fewer Black women experience IPV-related Post Traumatic Stress Disorder symptoms compared to White women, though they are also less likely to seek help from healthcare organizations.

IPV impacts HIV care engagement among Black women LWH. Attending HIV care visits is a critical step to HIV care engagement because interactions with healthcare providers can increase access to life-preserving antiretroviral therapies and other resources to address IPV. However, Black women experiencing various types of IPV (psychological, physical, and sexual) are less likely to access HIV healthcare. Among women already engaged in healthcare, women experiencing IPV are also more likely to experience hospitalizations and longer care disruptions compared to women not experiencing IPV. Thus, Black women LWH have increased risks of clinical progression if IPV is a barrier to full HIV care engagement. Barriers to HIV visit attendance reported among individuals experiencing IPV in previous studies have included: psychological control of money and/or resources by abusive partners, fear of rejection or escalated violence in response to disclosure of HIV status, overall poor health, low self-esteem, low self-efficacy, and fears of stigma.

The effects of stigma on HIV care engagement are pervasive among women experiencing HIV and IPV. The intersection of two socially devalued identities, HIV diagnosis and experiencing IPV, can cause psychological and emotional distress among BWLWHI. Factors driving stigmatization include societal beliefs that delegitimize BWLWHI, internalization of those beliefs, and fears about possible rejection if others know about their HIV status and IPV experiences. A recent systematic review found HIV-related stigma at multiple levels the most prevalent barrier to engaging in HIV care among Black women LWH. IPV stigma is a barrier to engaging with familial or friend networks for social support due to beliefs that women in violent relationships are irresponsible and unwise. Both of these societal stigmas are pervasive, and can affect individual decisions to employ IPV safety strategies and engage in HIV care.

Black women use IPV safety strategies and build on existing sources of strength to overcome the effects of IPV and HIV. Several studies report Black women LWH and/or experiencing IPV draw on internal and external sources of strength and employ safety strategies to overcome stigmas and preserve or improve their health. Women experiencing IPV reported accessing sources of strength to gain motivation to change their situation, leave their abuser, or take care of their health. Internal sources of strength include spirituality/religion or belief in God and self-reliance or belief in oneself. External sources included accessing informal and formal resources for support. Examples of informal support resources included friends or family who cared about the woman. Among Black women LWH, social support from family members, friends, and peers were resources for resilience; fostering health promoting behaviors to cope with HIV. Formal support resources for Black women experiencing IPV were police or court systems, IPV organizations, and healthcare. Feelings of empowerment and resiliency derived from a shared identity, unique strategies for coping, and awareness of social and political meaning can preserve Black women's well-being in the face of adversity. Black women LWH identified healthcare providers as vital resources of resilience to maintaining health. Resilience is linked to higher quality of life, undetectable viral load, and improved medication adherence among this group. Identifying the numerous ways women cope with IPV and build on their existing capacities are characteristics of strengths-based intervention approaches using a resiliency-reintegration model.

Strengths-based approaches engaging BWLWHI in care are lacking. Despite established links between IPV experiences and HIV care disengagement, few existing HIV care engagement interventions are tailored for Black women LWH nor do they address the effects of IPV on health. In fact, the majority of existing studies describe barriers and facilitators to care engagement but are not focused on interventions addressing these issues. The Living in the Face of Trauma (LIFT) intervention for women LWH found improved coping and reductions in traumatic stress 12 months after completing the intervention. However, this study did not focus on the role of current IPV. While strengths-based case management has been found to be a highly efficacious strategy to linking individuals to HIV care, it is resource-intensive and did not focus on the effects IPV can pose on this process. The negative influence of IPV experiences engagement in the distal outcomes of the HIV Care Continuum, i.e., medication adherence and viral suppression among Black women demonstrate potential areas for targeted intervention to address the effects of IPV and HIV-related stigma as barriers to HIV care visit attendance and receipt of ART.

The 1MoreStep study refines and tests a 8-session cognitive behavioral approach intervention referred to as COPE. COPE is a mnemonic of the skills: Challenge negative and maladaptive thoughts, Options - internal and external sources of strength, Positive affirmations, and Establish a plan. The investigators expect that introducing COPE skills will lead to increased HIV care engagement and use of IPV safety strategies in a sample of BWLWHI ages 18 and older.

The investigative team has a strong record of recruiting and retaining samples of Black women in Baltimore. The CHAT study (R01MH66810) was a Randomized Control Trial (RCT) testing a peer-based HIV prevention intervention with a sample of predominantly Black women. CHAT stands for: 1) Choose the right time and place; 2) Hear what the person is saying; 3) Ask Questions; and 4) Talk with respect. The Prevention and Testing study was a RCT testing an intervention for people LWH, 40% were Black women. The Young Women's Healthy Relationship (YWHR) study (R25-MH087217) was a cross-sectional study examining mental, sexual, and reproductive health effects of IPV and reproductive coercion among Black young women age 18 to 24 in Baltimore. The BMore PrEP Her Way (BHPHW) study (R24HD042854) recruited over 100 IPV-exposed women living in Baltimore to examine acceptability of women-controlled methods for HIV prevention (i.e. pre-exposure prophylaxis (PrEP)) and pregnancy prevention (long-acting reversible contraceptives (LARC)). Black women were 85% of the sample and 5% of the 250 screened ineligible were HIV-positive. Finally, myPlan, the IPV risk assessment and safety planning tool, that facilitators will introduce in Session 4 of the intervention was tested in diverse samples (>20% self-identified as Black women) and found to be an effective intervention for women experiencing IPV.

This study is a randomized, two-arm pilot clinical trial to determine acceptability, feasibility and preliminary estimates of efficacy of a trauma-informed cognitive behavior change program with 3-month and 6-month follow-up visits of BWLWHI (N=100). Participants complete baseline assessments and attend group sessions at a community-based research clinic. Follow-up assessments (satisfaction survey, qualitative interviews to assess acceptability and feasibility) will be conducted post-treatment and 3 and 6 months.

Experimental Condition: The intervention arm includes 7 small-group sessions and one individual session that meet weekly with facilitators who are paraprofessional women, one of whom is indigenous to the Black community in Baltimore and has experience implementing prior cognitive behavioral skills interventions in addition to several other HIV prevention and care RCTs with marginalized populations including Black women.

Session 1: The first session is an introduction of the purpose of the training and includes an activity about the strengths of BWLWHI and an inventory of internal and external sources of strength. Session 2: The intervention uses a mnemonic (COPE) to teach cognitive and behavioral skills, develop strategies for safety from IPV and improve knowledge and motivation for engagement in HIV care. Session 3: Teaches women about U=U and using COPE to address HIV care engagement. A female HIV care navigator will describe services offered at numerous clinics in Baltimore including the Baltimore Rapid Start Collaborative that provide immediate antiretroviral therapy to people newly diagnosed and/or re-engaging in HIV care. Participants will set HIV care goals. Sessions 4-5: These sessions are focused on conducting a personalized danger assessment and learning IPV safety strategies. In session 4, participants will meet in a small-group to learn about IPV safety strategies, specifically: placating strategies (e.g. not arguing with partner), safety planning (e.g. hiding car keys, keeping money hidden, having supplies ready for escape), engaging informal resources (e.g. sending kids to relatives) and formal resources (e.g. talking to a pastor, calling crisis line). Participants will be introduced to the myPlan app, which is a secure, interactive, and personalized app that has been developed and tested with diverse women (18 years and older) to support decisions to increase safety and reduce barriers to services. The myPlan app allows users to define their personal safety priorities, assess the level of danger in their intimate or dating relationship, and formulates a personally-tailored safety plan with referrals to appropriate resources and services. For the proposed study, no data will be used from the app. The app is a resource that will be shared with participants who are interested in voluntarily using it. The group will practice communication strategies for responding to enacted stigma which include positive affirmations such as "I am a survivor and doing the best I can for me and my kids", "One of my goals is to stay healthy for my kids, so going to the doctor is part of my plan", "I am worthy, HIV does not define me". Session 5 is an individual format in which the participant will identify the IPV safety strategies that she is willing to try and goal setting for safety planning. Session 6: The facilitator will discuss peer engagement, community building, and ways to support other Black Women Living With HIV (BLWHI). Session 7: This session is focused on goal setting for the next 30 days and establishing cues to remind the participant to practice the COPE skills. Session 8: Reunion session 30 days post completion of the intervention.

Comparison Condition: The Equal Attention Control/Standard of care control arm will consist of 7 group-based sessions that meet weekly and last 60-90 minutes. The control sessions provide both equal attention and psychotherapeutic experience of a support group where participants can talk about issues that are important in their lives, improving equal retention by study arm.

Session 1 will include a video entitled "Personal stories of people living with HIV" created by the Positive Life Campaign. Participants will share their experiences living with HIV and staff will give HIV care resources. Session 2 will be a standard of care presentation of IPV resources, services, and shelters for women. Sessions 3-5 will address diet-related health disparities that affect Black women such as obesity, hypertension and diabetes. Women will watch videos about each topic and then discuss their reactions. Session 6 will address caregiving and its relationship to self-care. Session 7 will address COVID-19 (transmission risks, symptoms and prevention behaviors) and related services available including food resources, financial assistance, testing sites and childcare. The investigators chose these topics because they are relevant to BWLWHI but not associated with the health outcomes targeted by the intervention.

Follow-up Assessments: All participants will be asked to complete a survey at 3 and 6 months post baseline. The follow-up surveys will assess changes in IPV safety strategies and HIV care linkage. Two participants per cohort will be asked to conduct an in-depth feedback interview.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender female
* Black or African American
* ≥ Age 18
* Living with HIV
* ≤ 1 HIV care visit in previous 12 months OR virally unsuppressed (>50 copies/mL) OR at high risk for poor HIV care adherence (PHQ ≥ 3, Generalized Anxiety Disorder (GAD) ≥ 3, active substance use)
* IPV within the previous 2 years
* Ability to attend in-person for up to 8 sessions
* Do not report immediate severe danger from their partner
* English fluency

Exclusion Criteria:

* Not a Cis-gender female
* Not Black or African American
* ≤ Age17 or younger
* Not living with HIV
* ≥ 2 HIV care visits in previous 12 months
* No IPV within the previous 2 years
* Inability to attend in-person for up to 8 sessions
* Reports immediate severe danger from their partner
* Not fluent in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as "cisgender": a cisgender woman is a person who was assigned female at birth and presents as a woman
Enrollment: 100 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Acceptability of study as measured by the Treatment Acceptance Scale | Week 7
  This scale has scores that range from 8 to 40. Low acceptability scores will be between 8 and 24, and high acceptability scores will be between 17 and 40.
Acceptability of study as measured by the Treatment Acceptance Scale | 3 month follow up
  This scale has scores that range from 8 to 40. Low acceptability scores will be between 8 and 24, and high acceptability scores will be between 17 and 40.
Acceptability of study as documented in in-depth interviews | 3 month follow up
  Interviews will assess program fit, facilitators and barriers to participation, and use of 1MoreStep intervention skills.
Feasibility of study as measured by session attendance | Week 7
  Session attendance

SECONDARY OUTCOMES:
Change in Intimate Partner Violence safety strategies as measured by the Intimate Partner Violence Safety Strategies Index | Baseline, Week 7 and 3 month follow up
  Four subscale scores will be evaluated independent of one another: accessing formal resources; accessing informal resources; placating strategies; and safety planning. Scores can range from a minimum of 0 to a maximum of 28. Scores which increase >1 in magnitude from baseline will indicate increased use of Intimate Partner Violence safety strategies by the participant, and therefore would be a positive outcome.
Change in Self-reported HIV Care Engagement in the form of ART medication use | Baseline, Week 7 and 3 month follow up
  Self-reported use of ART medication (yes or no)
Change in Use of prescription ART medication as assessed by chart review of HIV Care Engagement | Baseline, 3 month follow up and 1 year
  Chart review regarding use of prescription ART medication (yes or no)
Change in Number of HIV Care Provider visits as assessed by self-reported HIV Care Engagement | Baseline, Week 7 and 3 month follow up
  Self-reported HIV Care Engagement in the form of number of HIV Care Provider visits within the last year.
Change in Number of HIV Care Provider visits as assessed by Chart review of HIV Care Engagement | Baseline, 3 month follow up and 1 year
  Chart review regarding HIV Care Engagement in the form of HIV Care Provider visits within the last year.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Alexander, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Background] Turan B, Hatcher AM, Weiser SD, Johnson MO, Rice WS, Turan JM. Framing Mechanisms Linking HIV-Related Stigma, Adherence to Treatment, and Health Outcomes. Am J Public Health. 2017 Jun;107(6):863-869. doi: 10.2105/AJPH.2017.303744. Epub 2017 Apr 20. PMID 28426316
- [Background] Sikkema KJ, Ranby KW, Meade CS, Hansen NB, Wilson PA, Kochman A. Reductions in traumatic stress following a coping intervention were mediated by decreases in avoidant coping for people living with HIV/AIDS and childhood sexual abuse. J Consult Clin Psychol. 2013 Apr;81(2):274-83. doi: 10.1037/a0030144. Epub 2012 Oct 1. PMID 23025248